CLINICAL TRIAL: NCT04755179
Title: The Identification of the Optimal Treatment Strategy for Complex Appendicitis in the Pediatric Population
Brief Title: Identification of the Optimal Treatment Strategy for Complex Appendicitis in the Pediatric Population
Acronym: CAPP
Status: Completed | Type: Observational
Sponsor: Ramon Gorter (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor-Investigator, Ramon Gorter, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W18_302#18.348
Record Dates: First submitted 2021-01-29; First posted 2021-02-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Appendicitis; Appendix Mass; Appendicitis Perforated
Keywords: Complex appendicitis; Children; Treatment
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complex appendicitis without abscess or mass formation: All children (<18 years old) that present with a suspicion of complex appendicitis without clinical or radiological signs of abscess or mass formation. Preoperative suspicion of complex appendicitis is based upon a previously developed clinical scoring system.
  Interventions: Procedure: Laparoscopic appendectomy; Procedure: Open appendectomy
- Complex appendicitis with abscess or mass formation: All children (<18 years old) that present with a suspicion of complex appendicitis with clinical or radiological signs of abscess or mass formation. Preoperative suspicion of complex appendicitis is based upon a previously developed clinical scoring system.
  Interventions: Procedure: Non-operative treatment; Procedure: Direct appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy is performed according to daily practice but with the following standardized key points:
  1. Conventional laparoscopy (three-trocar technique)
  2. In case of purulent fluid: Suction and no peritoneal lavage procedure
  3. Skelletizing of the mesoappendix (coagulation/clips according to routine practice locally)
  4. Appendiceal stump closure: with two endoloops and dissected between the endoloops. In case of involvement of the appendiceal base, the use of endostapler is recommended.
  5. Withdrawal of appendix: principle of abdominal wall protection is followed (trocar technique / endobag)
  6. No drain placement, no nasogastric tube, and no urinary catheter routinely, only on indication.
  7. Closure of wounds as appropriate
  Groups: Complex appendicitis without abscess or mass formation
Procedure: Open appendectomy — Open appendectomy will be performed according to the following standardized key points:
  1. Gridiron incision at the right lower quadrant. (McBurney's point)
  2. After obtaining access to the abdominal cavity the principle of abdominal wall protection will be followed.
  3. The appendiceal stump will be closed by ligation, not a purse string suture.
  4. Closure of wounds as appropriate
  Groups: Complex appendicitis without abscess or mass formation
Procedure: Non-operative treatment — Non-operative treatment consisting of administration of intravenous antibiotics with or without drainage procedures (in case of an abscess), reserving an appendectomy for those not responding or with recurrent disease.
  One of the two antibiotic regiments:
  1. Combination A:
     1. Amoxicillin/clavulanic acid 25/2.5mg/kg 6 hourly (total 100/10 mg/kg daily. Maximum 6000/600mg a day) for children <40 kg OR Amoxicillin/clavulanic acid 1000/200mg/kg 8 hourly (total 3000/6000 mg/kg daily) for children > 40 kg
     2. Gentamicin 7mg/kg once daily
  2. Combination B:
     1. Cefuroxim 25 mg/kg 6 hourly (total 100 mg/kg/day. Maximum 6gram/day)
     2. Metronidazole 10mg/kg 8hourly (total 30 mg/kg/day. Maximum 4000 mg/day) In case of peri-appendicular abscess the decision can be made to perform a drainage procedure either percutaneously or surgical.
  Groups: Complex appendicitis with abscess or mass formation
Procedure: Direct appendectomy — laparoscopic or open appendectomy as described
  Groups: Complex appendicitis with abscess or mass formation

SUMMARY:
Aim of this study is to evaluate the effect of different treatment strategies on overall complications, health related-Quality of Life (hr-QOL) and costs among two subtypes of complex appendicitis in children (<18 years old).

Main research questions: What is the difference in overall complications at three months between:

Subgroup 1 (complex appendicitis without abscess/mass formation): Laparoscopic (LA) and open appendectomy (OA) Subgroup 2: (complex appendicitis with abscess/mass formation): Non-operative treatment (NOT) and direct appendectomy

DETAILED DESCRIPTION:
Up till now initiated research projects worldwide mainly focus on simple appendicitis (questioning the necessity of an appendectomy). However, complex appendicitis is associated with significant morbidity (up to 30%), prolonged hospital stay and high costs. Identification of the optimal treatment strategy for children with complex appendicitis is therefore essential. Heterogeneity in the treatment of complex appendicitis still exists in daily practice and reflects the lack of high-quality data and emphasizes the need for well-designed studies. Complex appendicitis can be divided into two subtypes:

1. Complex appendicitis without mass/abscess. (subgroup 1) Although (inter)national guidelines agree that appendectomy should be usual care, the optimal approach (open or laparoscopy) is unclear. Laparoscopic appendectomy (LA) is increasingly applied both in adults (80%) and children (60%). Benefits reported for LA in children are, but not limited to, less superficial site infection (SSI), reduced length of hospital stay and significant less postoperative bowel obstruction compared with open appendectomy (OA). Reluctance for usage of LA in this specific subgroup, however, remains due to the potential higher incidence of post-appendectomy abscess formation (PAA) reported. However, the quality of studies on this topic is low and there is considerable inconsistency in results.
2. Complex appendicitis with mass/abscess. (subgroup 2) The recommendation made in our national guideline (to perform direct appendectomy in this subgroup) is not in line with the available literature. A recent Cochrane review on this topic could only include two trials and stated that no firm conclusions could be drawn. An older systematic review, including 7 studies in children, concluded that non-operative treatment (NOT) led to fewer complications, specifically SSI and PAA, when compared to direct appendectomy. Still the recommendation from our national guideline is to perform a direct appendectomy based upon good experiences in the pediatric academic centers.

In order to investigate the optimal treatment for children with complex appendicitis we will perform a nationwide, multi-center, comparative, prospective cohort study. For the purpose of this study, treatment strategies will be standardized among the participating hospitals in order to reduce heterogeneity. Prospectively derived, high quality data will be sufficient to answer the research questions regarding the optimal treatment strategy for each subtype of complex appendicitis in the pediatric population. As it is a non-randomized prospective cohort study, propensity score matching technique will be performed in order to estimate the effect of the treatments adjusted for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

Eligible for inclusion are all children <18 years old that need to undergo treatment for the suspicion of complex appendicitis. Suspicion of complex appendicitis is based upon the following predefined criteria:

4 or more points on our scoring system developed to predict complex appendicitis. The diagnostic accuracy of this scoring system is 91% (Range: 84-98%). This scoring system consists of five variables (clinical, biochemical and radiological,each awarded points). In case the total score is 4 or more points, the patient is likely to have complex appendicitis. Variables included in the scoring system are:

* Diffuse abdominal guarding (3 points)
* CRP level more than 38 mg/L (2 points)
* Signs on ultrasound / imaging indicative for complex appendicitis (2 points)
* More than one day abdominal pain (2 points)
* Temperature more than 37.5 degrees Celsius (1 point)

Or

High index of suspicion of complex appendicitis by the treating physician. If this is the case, the treating physician will make pre-treatment note upon what clinical, biochemical or radiological variable the high index of suspicion is based.

Exclusion Criteria:

* Adult patients (=18 years old)
* Children with a suspicion of simple appendicitis (based upon the previous mentioned scoring system and radiological features)

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children that present with a preoperative suspicion of complex appendicitis. This suspicion is based on 4 points or more on the abovementioned complex appendicitis scoring system OR a high index of suspicion of complex appendicitis by the treating physician.
Sampling Method: Probability Sample
Enrollment: 1308 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Overall complications | 3 months
  The proportion of patients experiencing any complication within 3 months after inclusion

SECONDARY OUTCOMES:
Postappendectomy abscess | 3 months
  Proportion patients with a postappendectomy abscess
Superficial Site Infection | 3 months
  Proportion of patients with a superficial site infection
Secondary bowel obstruction | 3 months
  Proportion of patients with a secondary/prolonged bowel obstruction
Days absent from school, social or sports events | 30 days, 3 months
  Number of days absent from school, social or sports events
Number of days absent from work | 30 days, 3 months
  Number of days that parents are absent from work
Total number of extra visits | 30 days, 3 months
  Total number of extra visits to the outpatient clinic, general pratctitioner's office or emergency department
Length of hospital stay | 3 months
  Total length of hospital stay during follow-up due to trategy related treatment or complications
Level of pain | at inclusion/baseline (=day 0), 3 days, 5 days, 30 days, 3 months
  Level of pain measured according to the Visual Analogue Scale (0-10 points, higher scores indicating worse outcomes)
Pain medication utilization | 30 days, 3 months
  Pain medication utilization during admission
Need for appendectomy | 3 months
  Proportion of patients not having to undergo appendectomy within 3 months after start of non-operative treatment
Recurrent appendicitis | 3 months
  Proportion of patients experiencing recurrent appendicitis within 3 months after inclusion
Early failure of non-operative treatment | 3 months
  Proportion of patients experiencing early failure of initial non-operative treatment
Quality of Life questionnaire (EQ-5d-Youth/EQ-5d-Proxy) | at inclusion/baseline (=day 0), 30 days, 3 months
  QoL measured by the validated EQ-5d-Youth / EQ-5d-Proxy questionnaire (0-1 point, higher scores indicating better outcome)
Quality of Life questionnaire (PedsQL 4.0) | at inclusion/baseline (=day 0), 30 days, 3 months
  QoL measured by the validated Pediatric Quality of Life Inventory 4.0 (PedsQL 4.0) (0-100 points, higher scores indicating better outcome) Labor Questionnaire (HLQ), Medical Consumption Questionnaire (iMCQ) and Productivity Consumption Questionnaire (iPCQ) and gathered actual health care cost
Medical costs (iMCQ) | at inclusion/baseline (=day 0), 30 days, 3 months
  Medical costs measured by the iMedical Consumption Questionnaire
Non-medical / indirect costs (iPCQ) | at inclusion/baseline (=day 0), 30 days, 3 months
  Non-medical / indirect costs measured by the iProductivity Cost Questionnaire
Quality adjusted life months (QALM's) | 3 months
  Quality adjusted life months calculated using outcomes 14 -17
Patient satisfaction questionnaire (PSQ-18) | 3 months
  Patient satisfaction measured by the Patient Satisfaction Questionnaire (PSQ) (0-100, higher scores indicating better outcome)
Patient satisfaction questionnaire (Net promotor score) | 3 months
  Patient satisfaction measured by the NET PROMOTOR SCORE (0-10, higher scores indicating better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Gorter, MD PhD, Principal Investigator — Amsterdam UMC
Locations (32):
- Netherlands (32):
  - Northwest hospital group, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander MC, Amersfoort
  - Hospital Amstelland, Amstelveen
  - Amsterdam UMC - Location AMC, Amsterdam
  - Amsterdam UMC - Location VUmc, Amsterdam
  - OLVG, Amsterdam
  - Gelre hospital, Apeldoorn
  - Rijnstate, Arnhem
  - Bravis Hospital, Bergen op Zoom
  - Red Cross Hospital, Beverwijk
  - Tergooi, Blaricum
  - Amphia, Breda
  - IJsselland Hospital, Capelle aan den IJssel
  - Albert Schweitzer Hospital, Dordrecht
  - Catharina hospital, Eindhoven
  - Admiraal de Ruyter Hospital, Goes
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - Zuyderland MC, Heerlen
  - Dijklander, Hoorn
  - Sint Antonius Hospital, Nieuwegein
  - Radboud UMC, Nijmegen
  - Laurentius, Roermond
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Haga/JKZ, The Hague
  - Maxima Medical Centre, Veldhoven
  - Zaans Medical Centre, Zaandam
  - Isala, Zwolle

REFERENCES:
- [Derived] van Amstel P, Bakx R, van der Lee JH, van der Weide MC, Eekelen RV, Derikx JPM, van Heurn ELW, Gorter RR; CAPP collaborative study group. Identification of the optimal treatment strategy for complex appendicitis in the paediatric population: a protocol for a multicentre prospective cohort study (CAPP study). BMJ Open. 2022 Feb 17;12(2):e054826. doi: 10.1136/bmjopen-2021-054826. PMID 35177453